CLINICAL TRIAL: NCT03681041
Title: Pancreatic Injury and Corresponding Management Outcome (PICO): Prospective Multicenter Cohort Study From the Tertiary Referral or University-affiliated Hospitals
Brief Title: Pancreatic Injury and Corresponding Management Outcome (PICO)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Clinical Professor, Nanjing PLA General Hospital
Other Study IDs: 2021DZGZR-YBB-009
Record Dates: First submitted 2018-09-13; First posted 2018-09-21 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Trauma
Keywords: Pancreatic injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples analyses are performed by dedicated research center: DNA, and RNA extraction for transcriptome analysis, histological analyzes, etc: The concentrations of cell-free DNA, cell-free nucleosomes, neutrophil elastase (NE) and myeloperoxidase (MPO) were measured in sera and plasma by Human Cell Death Detection ELISA or sandwich ELISA.
  Pancreatic tissue was removed rapidly and divided into different parts for later analyses. One was used for confocal microscopy and one third was snap-frozen in liquid nitrogen for biochemical quantification of pancreatic myeloperoxidase (MPO), histone 3, and histone 4 levels, etc. One was fixed in formalin for histologic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic injury: Patient diagnosed with pancreatic trauma by surgery, computed tomography, Endoscopic retrograde cholangiopancreatography (ERCP) and Magnetic resonance cholangiopancreatography (MRCP) were included
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Standard treatment — Treatment according to guidelines for pancreatic trauma according to the Chinese Trauma Association and the American Association for the Surgery of Trauma

SUMMARY:
Pancreatic injury is a relatively rare and result in significant morbidity and mortality.

Estimates for the incidence of pancreatic injury range from 0.2-12% of abdominal traumas. Many factors, such as patient stability, the acuity of concomitant life-threatening injuries, and the need for damage control procedures must therefore be balanced when considering the proper approach to pancreatic injury management.

However, few prospective studies have investigated the perioperative management of patients with pancreatic trauma.

DETAILED DESCRIPTION:
Pancreatic trauma, while uncommon, presents challenging diagnostic and therapeutic dilemmas to trauma surgeons. Indeed, injuries to the pancreas have been associated with reported morbidity rates approaching 45%.

The disease 's characterization at a specific therapeutic level will allow for a better management of patients treated. To do so, the strategy is to integrate precise prospective clinical records extensive clinical treatment data in a large cohort of patients.

All the clinical departments, participating in the study, include patients, with a tight collaboration between Trauma, Intensive Care and Surgery departments. Demographics and clinical parameters are collected in a database.

Once after the diagnosis is confirmed, the inclusion of patients is performed, before a scheduled hospital management, and after eligibility criteria checking, and consent form signature. During clinical management, several samples are collected: blood samples and surgical specimens. As usual practice, post-operative treatment will be prescribed at investigator's discretion, with help of a pre-established algorithm. Several samples are also collected during this exam (blood and biological tissue sample).

At the same time as these managements, clinical data regarding medical history, pre-hospital treatment history, surgical history, treatments history, post-operative treatment if prescribed, treatments history between surgery and imageological diagnosis are recorded. Clinical data are also collected 12 months after discharge during a scheduled visit organized as usual practice, for long-term study.

Several studies will be performed along the cohort setting-up:

* Comparison of operative and non-operative treatment of pancreatic trauma:
* Comparison of the diagnosis time and treatment time of patients with pancreatic trauma and whether or not the treatment is missed
* Study of specific treatment of patients with pancreatic trauma
* Study of surgical methods and intraoperative conditions in patients with pancreatic trauma
* Study of ICU resuscitation treatment of patients with pancreatic trauma
* Study of endoscopy and other conservative treatments for patients with pancreatic trauma
* Study of nutritional support treatment for patients with pancreatic trauma
* Study of treatment methods for damage control and non-damage control in patients with severe pancreatic trauma

All the biologic samples are stored on sites at -80°C, or at room temperature depending on the samples: Samples collected in tubes, are sent immediately, at room temperature, to the central pathology department in Jinling Hospital, Nanjing, China. All the other samples, stored at -80°C, are sent to the Research Institute of General Surgery, Medical School of Nanjing University, China.

Samples analyses are performed by dedicated research center: DNA, and RNA extraction for transcriptome analysis, histological analyzes, etc:

Histological analyzes: Analysis of the structure of the excised pancreas or intestinal tissue.

Molecular Biology: Whole genome expression analyses are performed using microarray and followed by Gene Ontology and clustering analyses.

Microbiota: Bacterial composition of the ileal mucosa-associated microbiota is analyzed at the time of surgery using 16S (MiSeq, Illumina) sequencing. The obtained sequences are analyzed using the Qiime pipeline to assess composition, alpha and beta diversity.

Immunology: Phenotype of immune cells: Immune cells are extracted from blood and fresh mucosal tissues. The phenotype of these cells is analyzed by cytometry.

Analysis of neutrophil extracellular traps:

The concentrations of cell-free DNA, cell-free nucleosomes, neutrophil elastase (NE) and myeloperoxidase (MPO) were measured in sera and plasma by Human Cell Death Detection ELISA or sandwich ELISA.

Pancreatic tissue was removed rapidly and divided into different parts for later analyses. One was used for confocal microscopy and one third was snap-frozen in liquid nitrogen for biochemical quantification of pancreatic myeloperoxidase (MPO), histone 3, and histone 4 levels, etc. One was fixed in formalin for histologic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with pancreatic trauma by surgery
* computed tomography
* Endoscopic retrograde cholangiopancreatography (ERCP)
* Magnetic resonance cholangiopancreatography (MRCP)

Exclusion Criteria:

* The patient underwent chemotherapies or radiotherapy
* immune system disease
* end-stage chronic organ failure
* moribund cases with multiple severe injuries
* died within 24 h of admission
* younger than 18 years
* pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were treated for pancreatic injuries at the Trauma Centres
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  All cause mortality within 30 days

SECONDARY OUTCOMES:
pancreatic associated complications | Through study completion, an average of 1 year
  Complications due to pancreatic problems
Non-pancreatic associated complications | Through study completion, an average of 1 year
  Abdominal complications of non-pancreatic problems
Organ failure | 30 days
  Organ failure caused by organ dysfunction
Systematic complication | 30 days
  Complications such as pneumonia, abdominal sepsis, etc
Operational intervention | 30 days
  Complications after treatment for patients require operational intervention
Days on total parenteral nutrition | Through study completion, an average of 6 months
  Treatment time of parenteral nutrition support required during hospitalization
Time to enteral nutrition | Through study completion, an average of 6 months
  Time from management to initiate enteral nutrition in pancreatic injury patients
Days to clear liquids | Through study completion, an average of 6 months
  The time when the drainage tube is pulled out after the patient's abdominal liquids cleated
Days to regular diet | Through study completion, an average of 6 months
  The time from the treatment to the normal eating of patients with pancreatic trauma
Postoperative 30-day adverse effects | 30 day
  All cause adverse effects within 30 days
Hospital length of stay | Through study completion, an average of 6 months
  Length of hospital stay
Intensive Care Unit length of stay | Through study completion, an average of 6 months
  Length of Intensive Care Unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Ding, MD, Study Director — Medical School of Nanjing University
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang K, Li K, Deng Y, Wang X, Yang C, Chu C, Li W, Li J, Ding W. Postoperative hemorrhage following pancreatic injury: Risk factors and clinical outcomes. J Hepatobiliary Pancreat Sci. 2023 May;30(5):644-654. doi: 10.1002/jhbp.1251. Epub 2022 Nov 3. PMID 36270802